CLINICAL TRIAL: NCT06773429
Title: Estradiol's Effect on Brain Age
Brief Title: Estradiol and Brain Age
Status: Completed | Type: Observational
Sponsor: International Research Training Group 2804 (Other)
Collaborators: University Hospital Tübingen (Unknown); DFG - Deutsche Forschungs Gemeinschaft (German Research Foundation) (Unknown); Mini Research Training Group (MRTG) (Unknown)
Responsible Party: Sponsor
Other Study IDs: E2BrainAge
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Estradiol (E2) Vs. Placebo (PLAC); Estradiol
Keywords: Neuroprotection; brain-age; neuroimaging; menstrual cycle; sex hormones; estradiol; women's mental health

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Naturally cycling women: Naturally cycling women during the early follicular menstrual cycle phase
  Interventions: Drug: E2 Valerate; Drug: Placebo

INTERVENTIONS:
Drug: E2 Valerate — To experimentally elevate E2 levels females received 6mg of E2 valerate (Progynova21©) on two consecutive days (in total 12mg).
Drug: Placebo — Placebo pills (blue-colored hard gelatine capsules filled with a mixture of 99.5% mannitol and 0.5% Aerosil (fumed silica)) have been administered for the placebo-controlled condition.

SUMMARY:
The ovarian hormone estradiol (E2) is suspected to have a neuroprotective effect on the brain. Further, it is associated with mental health and brain plasticity, function and connectivity. During the menstrual cycle, women experience fluctuation of E2. This is closely associate with neuroplasticity in regions with high estradiol receptor density, such as the hippocampus, anterior cingulate cortex, amygdala, hypothalamus, or the striatum. In the current study we are interested on the effects of E2 on the brain age, indicated by the comparison between the chronological age and the predicted brain age. In a double-blind within-subject study design, naturally cycling females during their follicular menstrual cycle phase (when their endogenous ovarian hormone levels are low) were either administered estradiol valerate (E2) or a placebo (PLAC) to rapidly increase E2 levels independent of other cycling ovarian hormones. Structural brain scans were assessed.

DETAILED DESCRIPTION:
In this project we assessed regularly cycling females in their early follicular menstrual cycle phase with/without experimentally elevated estradiol (E2) levels in order to examine E2's effect on the brain age. Thus, women were scanned twice in the MR-scanner (E2 vs. PLAC; separated by at least 2-3 months) to deduce underlying structural changes. E2 vs. PLAC were administered in a double-blind, counterbalanced, randomized order. E2 has been administered orally (in total 12mg; two doses à 6mg on two consecutive days). All participants additionally underwent a neuropsychological assessment (demographical data, psychological and clinical data: structured clinical interview, anxiety and depression traits, mood, verbal intelligence, cognitive flexibility, emotion regulation traits, self-esteem). Blood samples were taken to assess endogenous gonadal hormone levels before and after E2/PLAC intake.

ELIGIBILITY:
Inclusion Criteria:

* Biologically females (assigned sex at birth)
* Regular menstrual cycle lasting between 26 and 35 days
* Right-handedness

Exclusion Criteria:

* Present or past mental, neurological or endocrine disorders, neurological or head injuries
* Use of hormonal contraceptives during the last six months
* Any other medication intake including intake of antidepressants or neuroleptics
* Past and present pregnancies
* Contraindication for MRI such as:

  * People with non-removable metal objects on or in the body
  * Tattoos if not MRI-incompatible according to expert guidelines
  * Pathological hearing or increased sensitivity to loud noises
  * Claustrophobia
  * Surgery less than three months ago
  * Restricted vision

Ages: 19 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population mainly consists of residents of Tübingen and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Association between E2 administration and brain age | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration. Predicted brain age during the E2- and the PLAC-condition will be compared to the chronological age.
Association between E2 level and brain age. | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and corresponding hormone levels. Association of E2-level increase with the difference between the predicted brain age and the chronological age ("brain-age-gap", BAG) will be compared.

SECONDARY OUTCOMES:
Association between progesterone level and brain age. | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and corresponding hormone levels. Association of progesterone levels [nmol/l] with the BAG [years] will be assessed.
Association between testosterone level and brain age | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and corresponding hormone levels. Association of testosterone levels [nmol/l] with the BAG [years] will be assessed.
Association between subjective mood and brain age. | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and mood ratings. Association of mood ratings [Positive and negative affect PANAS, ratings from 1 to 5] with the BAG [years] will be assessed.
Association between depression scores and brain age | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and depression scores. Association of depression scores [Becks depression index BDI] with the BAG [years] will be assessed.
Association between anxiety scores and brain age | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and anxiety scores. Association of anxiety scores [State anxiety index STAI] with the BAG [years] will be assessed.
Association between self-esteem and brain age | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and self-esteem scores. Association of self-esteem scores [Rosenberg selfesteem] with the BAG [years] will be assessed.
Association between emotion-regulation and brain age. | Females were measured twice with at least two-three months apart; each time: approx. 10 minutes assessment of MRI-scans
  Assessed via anatomical MRI scans after E2 and PLAC administration and emotion-regulation scores. Association of emotion-regulation [Heidelberg form of emotion regulation HFRST and emotion regulation questionnaire ERQ] scores with the BAG [years] will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Derntl, Prof., Principal Investigator — Departement of Psychiatry & Psychotherapy
Locations (1):
- University of Tuebingen; Department of Psychiatry & Psychotherapy, Tübingen, Baden-Wurttemberg, Germany